CLINICAL TRIAL: NCT00609557
Title: A Single-Blind Placebo Run-in Study of Duloxetine for Activity-Limiting Osteoarthritis Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Mark D. Sullivan, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 04-3386-B01; F1J-MC-X007
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2008-02-07 (Estimated); Status verified 2008-01

CONDITIONS: Osteoarthritis; Pain
Keywords: osteoarthritis pain; activity limitation; antidepressant; depression; single-blind
MeSH Terms: conditions — Osteoarthritis; Pain; Depression | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): All subjects receive placebo for the first two weeks and then duloxetine for the next 10 weeks, but they are blind to what they are receiving.
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: duloxetine — Weeks 0-2 placebo Weeks 2-3 30mg duloxetine Weeks 3-4 60mg duloxetine Weeks 4-12 60-90mg duloxetine Week 13 30 mg duloxetine Week 14 stop

SUMMARY:
This will be a single-blind, placebo-run-in trial. Subjects will be informed that they may receive duloxetine or placebo during the course of the trial. All subjects will, in fact, receive placebo for the first two weeks. All subjects will then be placed on 60-90mg per day of duloxetine. Primary outcome assessment will compare pain intensity at 2 weeks (after placebo) to that at 12 weeks (after 10 weeks of duloxetine treatment).

Study Hypothesis:

In subjects who continue to have activity-limiting osteoarthritis pain after treatment with acetaminophen or non-steroidal anti-inflammatory agents, 60-90 mg Duloxetine per day over 10 weeks will provide significant additional pain relief over that achieved with placebo(> 30% reduction after Duloxetine treatment).

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80
* Physician diagnosis of OA in hip, knee or spine.
* Significant activity limitation due to pain for at least one month on the Western Ontario and McMasters University Osteoarthritis Index (WOMAC) and average pain >5/10 on Brief Pain Inventory despite adequate treatment with acetaminophen or NSAIDs. [This will identify an OA group with significant psychological distress and a desire for treatment.]
* Depression status is not restricted, but will be monitored with PRIME-MD interview and the SCL-20. We anticipate depressive symptoms will be common in this population due to the above requirement for activity limitation.

Exclusion Criteria:

* Cannot read and write English
* Significant cognitive impairment
* History of psychosis or mania
* Current suicidal ideation

  * Current substance abuse or dependence
  * Current use of opioids or any antidepressant medication
  * Use of investigational drug within the past month

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Difference in average pain intensity on Brief Pain Inventory | between 2 weeks and 12 weeks
Difference in pain intensity on Western Ontario McMasters University Osteoarthritis Index (WOMAC) | Difference between 2 weeks and 12 weeks

SECONDARY OUTCOMES:
Difference in pain interference on Western Ontario McMasters University Osteoarthritis Index (WOMAC) | Difference between 2 and 12 weeks
Difference in role function as assessed by the Sheehan Disability Scales | Difference between 2 and 12 weeks
Difference on observed physical function as assessed by the Aggregated Locomotor Function score | Difference between 2 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Sullivan, M.D., Ph.D., Principal Investigator — University of Washington